CLINICAL TRIAL: NCT05992077
Title: Pilot Therapeutic Study of DAA Treatment for Children and Adolescents With Active HCV Infection in Cambodia
Brief Title: Study of DAA Treatment for Children and Adolescents With Active HCV Infection in Cambodia
Acronym: HEPEDIAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institute Pasteur, Cambodia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12420 HEPEDIAC
Record Dates: First submitted 2023-06-28; First posted 2023-08-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Intervention Model Description: Non-comparative multicenter pilot therapeutic prospective study. First, all children aged ≥ 6 years old and adolescents (expected 21000 participants) will be screened for HCV infection using HCV rapid test. HCV RNA will be performed in case of HCV rapid test positivity. Then, children and adolescents confirmed with active HCV infection (positive HCV RNA) during the screening phase will be referred to a specific consultation for treatment after evaluation of liver disease. We expect to enroll 60 participants in the therapeutic phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic phase (Experimental): Children and adolescents confirmed with active HCV infection (positive HCV RNA) during the screening phase will be referred to a specific consultation in Kantha Bopha hospital in Phnom Penh, Jayavarman VII hospital in Siem Reap, National Pediatric Hospital and Battambang provincial hospital for treatment after evaluation of liver disease. Patients with a weight > 25 kg will be treated with a sofosbuvir/daclatasvir combination for 12 weeks with adult dose (400/60 mg), children with a weight between 14 and 25 kg will be treated with the same sofosbuvir/daclatasvir combination with the half adult dose (200/30 mg) for 12 weeks. For all children and adolescents, residual plasma concentrations (trough concentrations) of the drugs will be assessed after 2 weeks of treatment.
  Interventions: Drug: Sofosbuvir/Daclatasvir

INTERVENTIONS:
Drug: Sofosbuvir/Daclatasvir — Patients with a weight > 25 kg will be treated with a sofosbuvir/daclatasvir combination for 12 weeks with adult dose (400/60 mg), children with a weight between 14 and 25 kg will be treated with the same sofosbuvir/daclatasvir combination with the half adult dose (200/30 mg) for 12 weeks.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of sofosbuvir/daclatasvir combination for children aged ≥ 6 years old and adolescents with active HCV infection in Cambodia

DETAILED DESCRIPTION:
Non-comparative multicenter pilot therapeutic prospective study conducted in Phnom Penh, Siem Reap and Battambang province and divided in 2 phases:

Screening phase:

First, all children aged more than 6 years old and adolescents under 18 years old will be screened for HCV infection using Bioline HCV rapid test in several pediatric populations in Phnom Penh, Siem Reap and Battambang including children born from HIV/HCV co-infected women followed in OI/ART sites or born from HCV mono-infected women.

HCV RNA will be performed in case of HCV rapid test positivity. A case-control study will be performed to evaluate the risk factors associated to HCV acquisition. Cases will be defined as children with positive HCV RDT and controls as children with negative HCV RDT. Four controls will be randomly selected for one case.

Therapeutic phase:

Children and adolescents confirmed with active HCV infection (positive HCV RNA) during the first phase will be referred to a specific consultation in Kantha Bopha hospital in Phnom Penh, Jayavarman VII hospital in Siem Reap, National Pediatric Hospital and Battambang provincial hospital for treatment after evaluation of liver disease. Patients with a weight > 25 kg will be treated with a sofosbuvir/daclatasvir combination for 12 weeks with adult dose (400/60 mg), children with a weight between 14 and 25 kg will be treated with the same sofosbuvir/daclatasvir combination with the half adult dose (200/30 mg) for 12 weeks. For all children and adolescents, residual plasma concentrations (trough concentrations) of the drugs will be assessed after 2 weeks of treatment. For the first 20 children and adolescents included (10 children weighing between 14 and 25 kg and 10 weighing more than 25 kg), whatever their HIV status and ARV treatment, a complete pharmacokinetic analysis will be performed prior to drug administration and +1h, +2h, +6h and +10h after drugs intake. A non-compartimental analysis using Phoenix WinNonlin 8.1 (Certara, Princeton, NJ, USA) will be performed to estimate the pharmacokinetic parameters of sofosbuvir, GS-331007 and daclatasvir. Maximal concentration (Cmax), trough concentration at steady state (Ct), minimal concentration (Cmin) and the time required to reach Cmax (Tmax) are the observed parameters. The area under the curve (AUCtau) will be estimated by the linear up log down trapezoidal method using the predose concentration as 24-hour postdose concentrations.

ELIGIBILITY:
Inclusion Criteria:

Screening phase Inclusion criteria

* Aged ≥ 6 years old with weight ≥ 14 kg
* Aged <18 years old
* Informed consent obtained with information sheet given and explained before the inclusion visit, the consent form signed by at least one of the 2 parents or legal guardians and oral assent collected if the child ≥ 13 years old, at the latest the day of the inclusion

Non-inclusion criteria

- Any concomitant medical condition that, according to the clinical site investigator, would contraindicate the HCV screening

Therapeutic phase Inclusion criteria

* Aged ≥ 6 years old with weight ≥ 14 kg
* Aged < 18 years old
* HCV RNA detectable
* HCV treatment naive
* In case of HIV coinfection,

  * HIV-1 infection confirmed according to Cambodian screening policies
  * On ART for more than 6 months
  * CD4 cell-count> 100 cells/μL and > 15% and HIV viral load < 1000 copies/mL at inclusion visit
* Informed consent obtained with information sheet given and explained before the inclusion visit and the consent form signed by at least one of the 2 parents and oral assent collected if the child ≥ 13 years old, before any sample or drug administration corresponding to the therapeutic phase.

Non-inclusion Criteria:

* Suspicion of evidence of hepato-cellular carcinoma (HCC) or any other neoplasia
* Decompensated cirrhosis
* Co-infection with HBV (positive HBsAg)
* Advanced/terminal renal disease defined as serum creatinine clearance < 30 mL/min
* Active tuberculosis under treatment
* In case of HIV coinfection,

  * Repeated ART failures and impossibility of prescription of an effective ART regimen
  * Active opportunistic infection (OI)
* Current pregnancy or breast feeding
* Use of any drug known to interact with Sofosbuvir or Daclatasvir and for which temporary cessation or dose modification would be impossible
* Any concomitant medical condition that, according to the clinical site investigator, would contraindicate participation in the study
* Concurrent participation in any other clinical trial without written agreement of the two study investigators

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21000 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of sofosbuvir/daclatasvir combination for children aged ≥ 6 years old and adolescents with active HCV infection in Cambodia | 24 months
  The proportion of patients with sustained virologic response defined by HCV RNA below the lower limit of quantification range of the viral load (undetectable viral load) 12 weeks after discontinuation of study drugs (SVR12). Detectable HCV RNA at the SVR12 study visit, permanent discontinuation of DAA, death, discontinuation of the study (loss to follow-up, transfer-out) will be considered as failures.

SECONDARY OUTCOMES:
Evaluation of the liver-related events | 24 months
  * Proportion of patients with symptomatic cirrhosis and evaluation of Child-Pugh score
  * Median (IQR) of APRI score and proportion of patients with APRI (AST to Platelet Index Ratio) score > 1
  * Proportion of patients with liver elasticity > 8 kPa
  * Proportion of patients with hepato-cellular carcinoma (HCC)
Occurrence of grade 3-4 adverse events (ANRS grading table); | 24 months
  * Frequency, type and time to grade 3 or 4 adverse clinical or biological events. All adverse events will be graded according to the Division of AIDS ( DAIDS) grading table;
  * Frequency, type and time to drug-related clinical or biological adverse reactions of grade 3 or 4 or leading to treatment interruption
Adherence | 24 months
  The adherence to DAA treatment will be assessed by accountability (drug pill count)
Maximal Plasma Concentration (Cmax) of DAA | 24 months
  Cmax of Sofosbuvir, GS-331007 and Daclatasvir measured in plasma samples
Area under the plasma concentration versus time curve over the dosing interval (AUCtau) of DAA | 24 months
  AUCtau of Sofosbuvir, GS-331007 and Daclatasvir will be estimated by the linear up log down trapezoidal method

OTHER OUTCOMES:
Risk factors of HCV acquisition through questionnaire | 24 months
  Case-control study to evaluate the risk factors associated to HCV acquisition. The questionnaire include information on family disease history, medical care received (injections, blood transfusion, surgery), dental care, tatoos, injecting drug user, use of traditional medicine, and sharing of hygiene tools.

CONTACTS AND LOCATIONS:
Locations (4):
- Cambodia (4):
  - Battambang Provincial Hospital, Battambang
  - Kantha Bopha Hospital, Phnom Penh
  - National Pediatric Hospital, Phnom Penh
  - Jayavarman VII Hospital, Siem Reap

IPD SHARING:
Plan to Share IPD: Undecided